CLINICAL TRIAL: NCT06797206
Title: An Observational Study to Evaluate the Impact of Pregnancy and Parenthood in Females With Cystic Fibrosis and Their Offspring in the CFTR Modulator Era.
Brief Title: A Study of Females With CF Throughout Pregnancy and Post-partum, and Follow up of Their Offspring
Acronym: MATRIARCH_CF
Status: Recruiting | Type: Observational
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Collaborators: Cystic Fibrosis Trust (Other); King's College London (Other); Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 352398
Record Dates: First submitted 2025-01-16; First posted 2025-01-28 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Cystic Fibrosis (CF); Pregnancy; Infant, Newborn; Exposure During Pregnancy
Keywords: Pregnancy/obstetric health in women with cystic fibrosis; Pregnancy; CFTR modulators
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Sputum, serum and urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Mama: Females with Cystic Fibrosis who are pregnant or planning a pregnancy
- Mini: Children aged 0-24 months with one biological parent who has a diagnosis of cystic fibrosis
- Midi: Children aged 3-6 years with one biological parent who has a diagnosis of cystic fibrosis

SUMMARY:
In this study, investigators aim to study in detail the physical (including nutritional and pulmonary) and mental health of females with cystic fibrosis (CF) planning a pregnancy, during pregnancy, and in the early parenthood period.

Additionally the health of offspring in infancy and early life will be studied to understand if further screening investigations or clinical care models should be part of clinical guidelines

DETAILED DESCRIPTION:
Improvements in treatments for people with CF have meant that more are becoming pregnant. CFTR modulators (CFTRm) are one of these treatments. They work by tackling the underlying cause of CF. These changes have created a need and an opportunity for research into the health and experiences of people with CF and their children in the CFTRm era.

The study is called 'MATRIARCH_CF' and includes 3 related sub-studies:

'Mama' is enrolling participants aged 16 years or older with CF under the care of the Royal Brompton Hospital (RBH) adult CF Unit who are planning a pregnancy or pregnant. The aim is to describe the impact of pregnancy and the first 12-24 months of parenthood in females with CF on their physical and psychological health. Investigations in eight visits include blood tests, lung function, imaging, and interviews.

'Mini' is enrolling biological offspring of people with CF (mothers and fathers) cared for by the RBH Adult CF Service, from birth to age two. The aim is to collect information that will allow for assessment of health outcomes in offspring of parents with CF in the short term. There will be up to four visits over two years with investigations including blood tests, sweat tests, and brain ultrasound.

'Midi' explores the same question as 'Mini' but in the longer term for those aged three-to-six. There will be up to two visits, and they include lung function testing and a lung MRI.

This study is described as 'observational' as investigators will not provide or change any treatment. Participant's health will be monitored with a range of investigations, many of which are optional. Knowledge gained from this study will be used to create guidelines to help families with CF and their medical teams make decisions around pregnancy and their offspring.

ELIGIBILITY:
Inclusion Criteria:

'Mama' sub-study:

* Written informed consent obtained from participant.
* Under the care of Royal Brompton Hospital CF Reproductive and Maternal Health Service
* Age 16 years or above at time of recruitment
* Confirmed diagnosis of CF
* Planning a pregnancy or pregnant at time of recruitment.
* Ability to adhere to the required visits and investigations.

'Mini' sub-study:

* Written informed consent obtained from participant's legal guardian.
* Infants who have one biological parent with a confirmed diagnosis of CF under care of Royal Brompton Hospital Adult CF Service
* Less than 12 months of age at first visit.
* Ability to adhere to the required visits and investigations.

'Midi' sub-study:

* Written informed consent obtained from participant's legal guardian.
* Children who have one biological parent with a confirmed diagnosis of CF who is under the care of Royal Brompton Hospital Adult CF Service.
* Age three to six years at time of visit
* Ability to adhere to the required visits and investigations.

Exclusion Criteria:

'Mama' sub-study:

* Any significant health condition which would cause inability to comply with protocol based on investigator discretion.
* History of lung transplantation

'Mini' sub-study:

* Legal guardians' inability to provide consent to participate in the study.
* Mother of infant has significant comorbidities unrelated to CF which could affect infant outcomes based on investigator discretion.

'Midi' sub-study:

* Legal guardians' inability to provide consent to participate in the study.
* A significant health condition which is known to affect lung function or imaging based on investigator discretion

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 1. Females aged 16 years or older with CF under the care of the Royal Brompton Hospital adult CF Unit who are planning a pregnancy or pregnant.
  2. Biological offspring of people with CF (both mothers and fathers) cared for by the Royal Brompton Hospital Adult CF Service, from birth to aged six years.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-06-12 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Change in FEV1 | 9 months
  Change in FEV1 percent predicted (ppFEV1) from pre-conception/baseline to end of pregnancy, and at 12- and 24-months post-partum.
Incidence of CF-related pulmonary complications during pregnancy. | 9 months
Incidence of premature delivery | 3 years
  Defined as birth <37 weeks gestation.
Frequency of liver dysfunction in infants | 2 years
  Defined as ALT/AST/GGT/bilirubin above upper limit of normal using laboratory normal ranges. This is prospectively obtained in the 'Mini' sub-study, and retrospectively reviewed from medical records in the 'Midi' sub-study.
Incidence of congential abnormalities | 3 years
  Based on medical history and examination
Frequency of CF diagnoses in infants despite negative newborn screen testing | 3 years
  The number of participants with normal IRT subsequently diagnosed with CF (based on a combination of CF genetic tests, sweat chloride, and faecal elastase where appropriate).
Frequency of abnormal lung clearance index results in young children | 3 years
  A lung clearance index (LCI) measurement above the normal levels as defined by investigating laboratory values (Midi only)

CONTACTS AND LOCATIONS:
Overall Officials: Imogen Felton, Principal Investigator — Royal Brompton Hospital and NHLI Imperial College London; Jane Davies, Principal Investigator — Royal Brompton Hospital and NHLI Imperial College London
Locations (1):
- Royal Brompton Hospital, London, United Kingdom